CLINICAL TRIAL: NCT03008629
Title: Clinical Efficacy of Nail Brace for Treatment of Ingrown Toenails
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Huang Yu Chen, Attending physician of Dermatology Department, Taipei Medical University WanFang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N201610005
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Ingrown Nail
MeSH Terms: conditions — Nails, Ingrown

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Podofix nail brace (Experimental): for mild ingrown toenails
  Interventions: Device: Podofix nail brace
- Combiped nail brace (Experimental): for Severe dystrophic ingrown toenails
  Interventions: Device: Combiped nail brace
- Podofix and then Combiped nail brace (Experimental): for Ingrown toenails with pyogenic granuloma
  Interventions: Device: Podofix and then Combiped nail brace

INTERVENTIONS:
Device: Podofix nail brace — Podofix nail brace
  Arms: Podofix nail brace
Device: Combiped nail brace — Combiped nail brace
  Arms: Combiped nail brace
Device: Podofix and then Combiped nail brace — Podofix and then Combiped nail brace
  Arms: Podofix and then Combiped nail brace

SUMMARY:
Background: Ingrown toenails are one of the most frequent nail disorders and can be treated with conservative or surgical approaches. Although discovered a long time ago, the available data are still very limited on the potential effectiveness of nail braces for ingrown toenail treatment.

Objective: This study aimed to evaluate the efficacy of nail brace (combiped and podofix) for treatment of ingrown toenails.

DETAILED DESCRIPTION:
Method: Participants with ingrown toenail and >= 12 years old with total 40 ingrown toenails were included. Investigators divide patients to 3 group: (1) combiped group: Participants with non-infected or mild infected ingrown nail, combiped nail brace was applied instantly.20 patients(2) combine combiped and podofix group: Participants with severe paronychia with pyogenic granuloma, oral analgesics and antibiotics were prescribed first and nail brace was applied 1 week later. Depends on disease condition, investigators applied 1-2 combiped nail brace. If the pyogenic granuloma is not resolved after 1 week, investigators applied podofix first for 2-4 weeks and then combiped nail brace. After the nail brace applied, participants must come back between 2-4 weeks depends on disease condition.10 patients (3) podofix group: participants who are afraid of combiped implantation, or with mild recurrence will be applied with podofix.

Participants come back every month for evaluation and photography. Physician global assessment (0-6),Patient global assessment (VAS 0-10), Treatment satisfaction (VAS 0-10), and questionnaire were evaluated 1 month, 3 months and 6 months after the device applied. Participants need to be followed for recurrence at 3rd month and 6th month after removed the nail brace.

ELIGIBILITY:
Inclusion Criteria:

* more or equal to 12 years old patient with ingrown toenail

Exclusion Criteria:

* < 12 years old
* under other nail bracing use
* received partial nail resection within recent 2 months
* psoriatic nail
* target therapy related paronychia
* received combiped or podofix previously and removed within recent 6 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Improvement (change) by Physician global assessment (0-6) | 1 month, 3 months and 6 months after the device applied

SECONDARY OUTCOMES:
Pain score (VAS0-10) | 1 month, 3 months and 6 months after the device applied
Improvement (change) by Patient global assessment (VAS 0-10) | 1 month, 3 months and 6 months after the device applied
Treatment satisfaction (VAS 0-10) | 1 month, 3 months and 6 months after the device applied
Quality of life by Questionnaire | 1 month, 3 months and 6 months after the device applied

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chen Huang, MD, Principal Investigator — Taipei Medical University WanFang Hospital

IPD SHARING:
Plan to Share IPD: No